CLINICAL TRIAL: NCT02081560
Title: Colistimethate and Colistin Pharmacokinetics in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy (CRRT)
Brief Title: Colistin Pharmacokinetics in Continuous Renal Replacement Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLPKZH11; 213DR11032 (Other: Swissmedic)
Record Dates: First submitted 2014-02-27; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Infection
Keywords: pharmacokinetics; antibiotic; Gram negative; continuous renal replacement therapy
MeSH Terms: conditions — Infections | interventions — Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- colistin pharmacokinetics (Other): Intravenous colistin 9 million units loading dose and 3 million units q8h maintenance dose as long as treatment of infection is required
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Colistin — Colistin i.v. three times daily as long a necessary for infection treatment

SUMMARY:
The blood concentration of the antibiotic colistin is determined in patients in whom kidney function is reduced such that a renal replacement therapy is needed.

Hypothesis:no dose reduction is needed in patients undergoing continuous renal replacement therapy over 24h because colistin is sufficiently removed by this procedure.

DETAILED DESCRIPTION:
After administration of intravenous Colistin multiple blood samples are drawn over one dosing interval on day 1, 3, and 5 of treatment.

Patients are monitored for signs of neuro- and nephrotoxicity

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18 years or older
* hospitalised on the ICU
* gram-negative infection requiring antibiotic therapy with intravenous colistin as part of their routine medical care
* clinical necessity for continuous venovenous renal replacement therapy

Exclusion Criteria:

* History of hypersensitivity to colistin or to other polymyxins
* Personal or family history of Myasthenia Gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) | predose, and 0.5, 1, 2, 4, 6, 8 hours after administration

SECONDARY OUTCOMES:
Sings of neurotoxicity and nephrotoxicity | Expected average of follow up is about 14 days.
  Clinical investigation daily by assessing clinical signs and questioning the patient regarding sign of neuropathy and difficulty breathing in non intubated patients. Questioning the treating physician in intubated patients regarding objective signs of increased ventilation support.
Sings of neurotoxicity and nephrotoxicity | Expected average of follow up is about 14 days.
  Clinical investigation daily by assessing clinical signs and questioning the patient regarding sign of neuropathy and difficulty breathing in non intubated patients. Questioning the treating physician in intubated patients regarding objective signs of increased ventilation support. The patients will be followed for the duration of colistin administration at the dose studied.

CONTACTS AND LOCATIONS:
Overall Officials: Natascia Corti, MD, Principal Investigator — University Hospital Zurich, Dept. of Pharmacology and Toxicology
Locations (1):
- University Hospital of Zurich, Dept. of Pharmacology and Toxicology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Leuppi-Taegtmeyer AB, Decosterd L, Osthoff M, Mueller NJ, Buclin T, Corti N. Multicenter Population Pharmacokinetic Study of Colistimethate Sodium and Colistin Dosed as in Normal Renal Function in Patients on Continuous Renal Replacement Therapy. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01957-18. doi: 10.1128/AAC.01957-18. Print 2019 Feb. PMID 30478168